CLINICAL TRIAL: NCT00704886
Title: A Randomized Controlled Trial of Using Video Images in Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Angelo Volandes, MD PI, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007p001264
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Dementia
Keywords: dementia
MeSH Terms: conditions — Dementia | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): verbal
- 2 (Experimental): video
  Interventions: Other: video

INTERVENTIONS:
Other: video — video of dementia
  Other Names: video decision aid
  Arms: 2

SUMMARY:
BACKGROUND: Advance care planning (ACP) is the process in which patients plan for future medical care under circumstances of impaired decision-making. Video is an underutilized medium that can assist clinicians in discussions of future health states, such as the state of advanced dementia. Video may enable patients to visualize the future by concisely providing complex information vital for ACP. This study will examine whether the use of video could facilitate a more comprehensive understanding of advanced dementia and inform clinician-patient discussions about the level of care a patient would want in the event of advanced dementia.

RESEARCH PLAN: We propose to conduct a randomized trial studying ACP for 200 elderly subjects using a video depiction of a patient with dementia compared to the traditional verbal narrative. Specific aims 1 and 2 assess the effect of a video of advanced dementia on the clinical decision making of elderly subjects compared to the traditional verbal narrative.

DETAILED DESCRIPTION:
Outcome measures were what subjects wanted if they had advanced dementia.

ELIGIBILITY:
Inclusion Criteria:

* Over 64

Exclusion Criteria:

* Can't speak English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
preferences | at time of interview

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, MD, Principal Investigator — MGH
Locations (1):
- MGH, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Volandes AE, Paasche-Orlow MK, Barry MJ, Gillick MR, Minaker KL, Chang Y, Cook EF, Abbo ED, El-Jawahri A, Mitchell SL. Video decision support tool for advance care planning in dementia: randomised controlled trial. BMJ. 2009 May 28;338:b2159. doi: 10.1136/bmj.b2159. PMID 19477893